CLINICAL TRIAL: NCT01267955
Title: A Phase 2 Study of GDC-0449 in Patients With Advanced Chondrosarcomas
Brief Title: Vismodegib in Treating Patients With Advanced Chondrosarcomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02564; NCI-2011-02564 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000691728; IB-CHONDROG; CHONDROG; 8408 (Other: Institut Bergonie Cancer Center); 8408 (Other: CTEP)
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Clear Cell Chondrosarcoma; Dedifferentiated Chondrosarcoma; Locally Advanced Chondrosarcoma; Mesenchymal Chondrosarcoma; Metastatic Chondrosarcoma; Primary Central Chondrosarcoma; Unresectable Primary Central Chondrosarcoma
MeSH Terms: conditions — Chondrosarcoma, Clear Cell; Chondrosarcoma, Mesenchymal; Chondrosarcoma | interventions — Pharmacogenomic Testing; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vismodegib) (Experimental): Patients receive vismodegib PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Drug: Vismodegib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC 0449; GDC-0449; GDC0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This phase II trial studies how well vismodegib works in treating patients with chondrosarcomas that have spread to other places in the body and usually cannot be cured or controlled with treatment. Drugs used in chemotherapy, such as vismodegib, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the antitumor activity of GDC-0449 (vismodegib) in terms of 6-month clinical benefit rate (complete response, partial response, and stable disease, as per the revised Response Evaluation Criteria in Solid Tumors [RECIST] criteria 2009).

SECONDARY OBJECTIVES:

I. Best overall response (as per the revised RECIST criteria 2009). II. 1- and 2-year progression-free survival. III. 1- and 2-year overall survival. IV. GDC-0449 safety. V. Pharmacogenomics analysis of predictive markers of treatment outcome.

OUTLINE:

Patients receive vismodegib orally (PO) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of chondrosarcoma (conventional, mesenchymal, dedifferentiated or clear cell subtypes)
* Patients must have measurable disease (outside any previously irradiated field) defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with spiral computed tomography (CT) scan
* No more than three prior lines of chemotherapy for advanced disease (including no more than 450 mg/m^2 doxorubicin); at least three weeks since last chemotherapy (six weeks in case of nitrosoureas and mitomycin C), immunotherapy or any other pharmacological treatment and/or radiotherapy
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Metastatic or unresectable locally advanced disease
* Documented disease progression (as per RECIST) before study entry
* Women of child-bearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 24 months post-treatment for female patients and for 2 months for male patients; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 7 days prior to initiation of GDC-0449 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks while on study within the 24-hour period prior to the administration of GDC-0449; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing GDC-0449, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of GDC-0449

  * Women of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had a tubal ligation
  * Women are considered not to be of childbearing potential for the following reasons:

    * The patient has undergone hysterectomy and/or bilateral oophorectomy
    * The patient is post-menopausal defined by amenorrhea for at least 1 year in a woman > 50 years old
    * The patient has permanent premature ovarian failure confirmed by specialist gynecologist
* Ability to understand and the willingness to sign a written informed consent document
* In accordance with French Regulatory Authorities: Patients with French Social Security in compliance with the French law relating to biomedical research (Huriet Law 88-1138 and related decrees)

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449 or other agents used in the study
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow capsules
* Patients with clinically important history of liver disease, including viral or other hepatitis, or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation, are excluded from this study
* Tumor tissue sample not available for pathological review and/or correlative studies
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with GDC-0449; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-12-21 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2026-07-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Italiano, Principal Investigator — Institut Bergonie Cancer Center
Locations (6):
- France (6):
  - Institut Bergonie Cancer Center, Bordeaux
  - Centre Oscar Lambert, Lille
  - Centre Leon Berard, Lyon
  - Hopital De La Timone, Marseille
  - Institut Curie Paris, Paris
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Italiano A, Le Cesne A, Bellera C, Piperno-Neumann S, Duffaud F, Penel N, Cassier P, Domont J, Takebe N, Kind M, Coindre JM, Blay JY, Bui B. GDC-0449 in patients with advanced chondrosarcomas: a French Sarcoma Group/US and French National Cancer Institute Single-Arm Phase II Collaborative Study. Ann Oncol. 2013 Nov;24(11):2922-6. doi: 10.1093/annonc/mdt391. PMID 24170610

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Vismodegib): Patients receive vismodegib PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacogenomic Study: Correlative studies
  Vismodegib: Given PO
  This is a single-arm phase 2 trial, based on a two-stage Simon's optimal design. Assuming 20% (H0: null hypothesis) and 40% (H1: alternative hypothesis) six-month CBR, 10% type I error rate and 90% power, 37 eligible and assessable patients were necessary (17 in the first stage and 20 in the second stage). At the second stage/final stage, GDC-0449 would be considered promising if at least eleven patients were progression-free at 6 months.
Period: Stage 1 (6 Months)
Arm/Group | Treatment (Vismodegib)
Started | 20
Completed (Subjects contributing data to the primary analysis are considered to have completed the study.) | 17
Not Completed | 3
Not completed — Death | 3
Period: Stage 2 (6 Months)
Arm/Group | Treatment (Vismodegib)
Started | 45
Completed | 39
Not Completed | 6
Not completed — Death | 5
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled
Arm/Group | Treatment (Vismodegib)
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 58.0 [27.0 to 85.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race and Ethnicity Not Collected Population: Race and Ethnicity Not Collected
Region of Enrollment [Number; unit: participants]
  France | 45
ECOG Performance status [Count of Participants; unit: Participants] — The ECOG scale of performance status developed by the Eastern Cooperative Oncology Group (ECOG) was used to assess the functional status of a patient in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). A grade 0 corresponds to a patient fully active, grade 1 a patient restricted in activity, grade 2 a patient capable of all selfcare but unable to carry out any work activities, grade 3 capable of only limited selfcare, grade 4 a patient completely disabled, grade 5 patient dead.
  Participants
    0 | 20
    1 | 20
    2 | 5
Weight [Median (Full Range); unit: kilogram] — Population: Weight not available for 1 patient
  kilogram
    number analyzed (Participants) | 44
    (all) | 76.5 [51.0 to 102.0]
Height [Median (Full Range); unit: millimetres] | 173.0 [148.0 to 200.0]
Histological subtype [Count of Participants; unit: Participants]
  Conventional chondrosarcoma | 39
  Dedifferentiated chondrosarcoma | 5
  Clear cell chondrosarcoma | 1
  Mesenchymal chondrosarcoma | 0
Stage of the disease [Count of Participants; unit: Participants]
  Locally advanced | 13
  Metastatic | 32
Prior lines of chemotherapy [Count of Participants; unit: Participants]
  0 | 25
  1 | 12
  2 | 3
  >2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) Based on Centralized Imaging Review as Per RECIST 1.1
Description: CBR was defined as the percentage of participants with complete or partial responses (CR, PR) or stable disease (SD) per RECIST 1.1. CR was defined as disappearance of all non-nodal target lesions. PR was defined as at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Analysis of response was performed based on radiological centralized review. A 2-stage optimal Simon's design with 37 participants (first stage: 17 participants) was used. If 3 or less non-progressions (CR + PR + SD) at 6 months were observed during stage 1 (out of 17 participants), the trial would stopped early. Otherwise, 20 additional patients would be accrued for stage 2. If 11 or more non-progressions (out of 37 participants) were observed at the end of recruitment, further investigation of this therapy would be warranted.
Time Frame: At 6 months after inclusion
Population: Eligible participants with at least one complete or two incomplete cycles of treatment and for whom at least one disease measurement has been recorded not less than 8 weeks after treatment onset.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Vismodegib)
Number analyzed (Participants) | 39
percentage of participants
  First stage: number analyzed (Participants) | 17
  First stage | 23.5 [6.8 to 49.9]
  Second stage (Overall) | 25.6 [13.0 to 42.1]

2. Secondary Outcome: Progression-free Survival
Description: Will be analyzed using the Kaplan-Meier method. The median survival rates will be reported with a 95% confidence interval. Median follow-up will be calculated using the reverse Kaplan-Meier method.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 3 years
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival Per Response Evaluation Criteria in Solid Tumors Criteria 2009
Description: Overall survival will be analyzed using the Kaplan-Meier method. The median survival rates will be reported with a 95% confidence interval. Median follow-up will be calculated using the reverse Kaplan-Meier method.
Time Frame: Time from start of treatment to the time of death, assessed up to 3 years
Reporting Status: Not Posted

4. Secondary Outcome: Duration of Response
Description: Will be described in responding subjects using descriptive statistics (median, extreme values, etc.).
Time Frame: From the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 3 years
Reporting Status: Not Posted

5. Secondary Outcome: Mutational Status of Patched 1 and Smoothened
Description: The 6-months clinical benefit rate will be correlated with the mutational status of patched and smoothened in order to identify predictive factors of clinical benefit from vismodegib.
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: Expression Pattern of Hedgehog Signaling Molecules by Using Quantitative Reverse Transcription-polymerase Chain Reaction and Immunohistochemistry
Description: The 6-months clinical benefit rate will be correlated with the expression score of hedgehog signaling molecules in order to identify predictive factors of clinical benefit from vismodegib.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 months of treatment. At the time of primary analysis, 8 were still on treatment and 37 patients discontinued treatment.
Description: Adverse event are reported for all treated patients who received at least one administration of treatment.
Arm/Group | Treatment (Vismodegib)
All-Cause Mortality (participants affected / at risk) | 23/45
Serious Adverse Events (participants affected / at risk) | 22/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vismodegib) (N=45)
ANEMIA (Blood and lymphatic system disorders) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2) — 2 patients with ALTERATION OF GENERAL STATUS;
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) — 1 patient with hepatic cytolysis
Sepsis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
GGT increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) — 3 patients with disease progression 1 patient with SPINAL CORD COMPRESSION 1 patient hospitalized for general status alteration
Cognitive disturbance (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (2) — 1 patient with TRANS TIBIAL AMPUTATION LEFT FOOT 1 patient with PARIECTOMY 7 TH, 8 TH AND 9 TH LEFT COAST + RESSECTION OF LUNG PARENCHYMA+ECCISION OF A NODULE PLEURAL
Thromboembolic event (Vascular disorders) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vismodegib) (N=45)
ANEMIA (Blood and lymphatic system disorders) | 9 (15)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 9 (9)
Constipation (Gastrointestinal disorders) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 13 (19)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 17 (20)
Stomach pain (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 7 (7)
Chills (General disorders) | 3 (4)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 24 (28)
Fever (General disorders) | 8 (13)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (3) — 1 patient with GENERAL STATUS IMPAIRMENT; 1 patient with GENERAL STATUS ALTERATION; 1 patient with GENERAL STATUS ALTERATION AND RIGHT UPPER LIMB DEFICIT
Bronchial infection (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 7 (9)
Alkaline phosphatase increased (Investigations) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 5 (5)
GGT increased (Investigations) | 5 (6)
Lymphocyte count decreased (Investigations) | 4 (5)
Weight loss (Investigations) | 12 (12)
Investigations - Other, specify (Investigations) | 5 (8) — 1 patient with LDH INCREASED; 1 patient with LACTATE DESHYDROGENASE INCREASED; 1 patient with LDH INCREASED; 1 patient with C PROTEIN REACTIVE INCREASED; 1 patient with INFLAMMATORY SYNDROME (WITH INCREASE OF CRP)
Anorexia (Metabolism and nutrition disorders) | 12 (15)
Hypercalcemia (Metabolism and nutrition disorders) | 7 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (9)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (6)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 23 (27)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) — 3 patients with disease progression; 1 patient with SPINAL CORD COMPRESSION
Dizziness (Nervous system disorders) | 3 (3)
Dysesthesia (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 29 (30)
Headache (Nervous system disorders) | 6 (8)
Paresthesia (Nervous system disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4)
Urinary frequency (Renal and urinary disorders) | 3 (21) — 1. patient with STOMACH PAIN; 2. patients with POLLAKIURIA
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (18)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) — 1 patient with RASH; 1 patient with DEPILATION; 1 patient with ANKLE BEDSORES
Lymphedema (Vascular disorders) | 3 (4)
Thromboembolic event (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT01267955/Prot_SAP_000.pdf